CLINICAL TRIAL: NCT05824832
Title: Effects of a Triple Adjuvant Combination of Buprenorphine, Clonidine, and Dexamethasone on Duration of Brachial Plexus Blocks for Upper Extremity Surgery, a Prospective, Randomized Clinical Trial
Brief Title: Buprenorphine, Clonidine, and Dexamethasone on Duration of Brachial Plexus Blocks for Upper Extremity Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Audrice Francois, MD, FASA, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 216009
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative
Keywords: buprenorphine; clonidine; dexamethasone; brachial plexus blocks; pain; shoulder; surgery
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Clonidine; Dexamethasone; Nerve Block; Buprenorphine

STUDY DESIGN:
Intervention Model Description: Prospective randomized single-blinded clinical trial. 1:1 Randomization with 2 groups.
  Group 1: 50% of participants will receive an Interscalene brachial plexus blocks with the addition of buprenorphine, dexamethasone, and clonidine during surgery.
  Group 2: 50% of participants will receive an Interscalene block alone during surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interscalene block with the addition of buprenorphine, clonidine, dexamethasone (Experimental): Interscalene brachial plexus blocks (ISB) is performed with a 22g x 50 mm PAJUNK SonoPlexⓇ II Facet S echogenic needle. Once adequate needle visualization is achieved within the correct anatomic position and plane, 30mL of 0.5% bupivacaine with 100 mcg clonidine, 0.3 mg buprenorphine, and 4 mg dexamethasone will be injected.
  Interventions: Drug: Interscalene block with the addition of buprenorphine, clonidine, dexamethasone
- Interscalene block with buprenorphine alone (Active Comparator): Interscalene brachial plexus blocks (ISB) is performed with a 22g x 50 mm PAJUNK SonoPlexⓇ II Facet S echogenic needle. Once adequate needle visualization is achieved within the correct anatomic position and plane 30mL of 0.5% bupivacaine will be injected.
  Interventions: Drug: Interscalene block with buprenorphine alone

INTERVENTIONS:
Drug: Interscalene block with the addition of buprenorphine, clonidine, dexamethasone — Addition of the adjuvant buprenorphine, dexamethasone, and clonidine in the nerve block performed prior to shoulder arthroscopy surgery
  Other Names: Nerve block with buprenorphine, clonidine, dexamethasone
  Arms: Interscalene block with the addition of buprenorphine, clonidine, dexamethasone
Drug: Interscalene block with buprenorphine alone — Addition of the adjuvant buprenorphine alone the in nerve block performed prior to shoulder arthroscopy surgery
  Other Names: Nerve block with buprenorphine alone
  Arms: Interscalene block with buprenorphine alone

SUMMARY:
The goal of this clinical trial is to learn if there is a difference in morphine requirements in patients after upper extremity surgeries including shoulder arthroscopy. The main question it aims to answer is whether there is a difference between Interscalene brachial plexus blocks with the addition of buprenorphine, dexamethasone, and clonidine and the same block without the adjuvant.

DETAILED DESCRIPTION:
This study will be a prospective randomized single-blinded clinical trial.

Patients undergoing shoulder arthroscopy who meet the inclusion criteria will be invited to participate in this study. A total of 120 patients will be recruited to participate.

Patients will be randomized via a 1:1 ratio to either the Interscalene block with the addition of buprenorphine, clonidine, dexamethasone group or Interscalene block alone group

The null hypothesis of this research study is that there will be no significant difference in morphine requirements between the Interscalene brachial plexus blocks with the addition of buprenorphine, dexamethasone, and clonidine and the same block without the adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Patients undergoing shoulder arthroscopy
* Patients willing to participate and sign informed consent

Exclusion Criteria:

* Severe COPD/other contraindication to general anesthesia
* Patient with a weight of less than 60 kg
* Dementia, not alert or oriented to person, place, or time
* Chronic pain patient with daily opioid use at home.
* Patient with allergy to local anesthetics
* Patient refusal
* Total shoulder arthroplasty
* Concomitant pain in different area from operative site.
* Pregnancy
* Patient with active infection on the injection sites for the blocks
* Patients unable or willing to understand or comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Morphine requirement post surgery | 24 hours
  To compare the morphine equivalents administered in the first 24 hours after arrival in the recovery area between the two groups.

SECONDARY OUTCOMES:
Pain reported via a numeric rating scale (NRS) | 48 hours
  To measure pain via a numeric rating scale (NRS) immediately after arrival to recovery area from surgery (time: 0hr), and again at 2, 24, and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Audrice Francois, MD, Principal Investigator — Loyola University Chicago
Locations (1):
- Loyola University Chicago, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No